CLINICAL TRIAL: NCT03251027
Title: Intensity-Modulated Stereotactic Radiotherapy as an Upfront Scalp-Sparing Intervention for the Treatment of Newly Diagnosed Grade II-IV Gliomas
Brief Title: Intensity-Modulated Stereotactic Radiation Therapy in Treating Patients With Grade II-IV Glioma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17D.074; JT 9581 (Other: JeffTrial Number)
Record Dates: First submitted 2017-08-14; First posted 2017-08-16 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Glioblastoma; WHO Grade II Glioma; WHO Grade III Glioma
MeSH Terms: conditions — Glioblastoma | interventions — Radiotherapy, Intensity-Modulated; Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (IM-SRT) (Experimental): Patients undergo intensity-modulated (IM)-stereotactic radiotherapy (SRT) daily over 6 weeks.
  Interventions: Radiation: Intensity-Modulated Radiation Therapy; Other: Quality-of-Life

INTERVENTIONS:
Radiation: Intensity-Modulated Radiation Therapy — Undergo IM-SRT
Other: Quality-of-Life — Ancillary studies
  Other Names: Quality of Life Assessment; Quality-of-Life Assessment

SUMMARY:
This phase II trial studies how well intensity-modulated stereotactic radiation therapy works in treating patients with grade II-IV glioma. Stereotactic radiosurgery is a specialized radiation therapy that delivers a single, high dose of radiation directly to the tumor and may cause less damage to normal tissue.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the effect of intensity-modulated (IM)-stereotactic radiotherapy (SRT) on the incidence of wound infection (requiring oral/intravenous [IV] antibiotics or surgery), or wound dehiscence.

SECONDARY OBJECTIVES:

I. To determine the effect of IM-SRT on the incidence of titanium implants as palpable cranial defects due to scalp thinning.

II. To determine the effect of IM-SRT on the incidence of hair loss and recovery rate.

III. To determine the effect on quality of life (QoL) using European Quality of Life Five Dimension Five Level Scale Questionnaire (EQ-5D-5L).

TERTIARY OBJECTIVES:

I. To determine if treatment of Intensity-modulated stereotactic radiotherapy (IM-SRT) in patients with newly diagnosed grade II-IV gliomas can decrease the loss of scalp thickness in the coronal plane in T-1W magnetic resonance (MR) images.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed low or high grade glioma (grade II-IV)
* Karnofsky performance status (KPS) >= 60
* Patients must have recovered from the effects of surgery; there must be a minimum of 21 days from the day of surgery to the day of protocol treatment
* Estimated survival >= 3 months
* Labs considered acceptable per standard of care
* Patient must sign a study specific informed consent form
* Radiation treatment must begin >= 3 weeks and =< 8 weeks after surgery

Exclusion Criteria:

* Prior history of scalp radiation or intolerance to standard course of radiation treatment
* Co-morbidities that would influence wound healing including diabetes (insulin dependent) or smoking (current ongoing use)
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception
* Karnofsky performance status (KPS) < 60
* Patient can't have magnetic resonance imaging (MRI) scan
* Active collagen vascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of wound infection or wound dehiscence | Up to 2 years
  Will assess the impact of intensity-modulated stereotactic radiotherapy (IM-SRT) on the incidence of wound infection, or wound dehiscence.

SECONDARY OUTCOMES:
Incidence of titanium implants | Up to 2 years
  Will the impact of IM-SRT on the incidence of titanium implants as palpable cranial defects due to scalp thinning. Rates of titanium implant discomfort will be summarized by cohort with exact 95% confidence intervals. Within-cohort changes will be estimated using linear contrasts of model parameters.
Incidence of hair loss | Up to 2 years
  Will assess the impact of IM-SRT on the incidence of hair loss. Will be summarized by cohort with exact 95% confidence intervals. Within-cohort changes will be estimated using linear contrasts of model parameters.
Incidence of recovery rate | Up to 2 years
  Will assess the impact of IM-SRT on the incidence of recovery rate. Will be summarized by cohort with exact 95% confidence intervals. Within-cohort changes will be estimated using linear contrasts of model parameters.
Quality of life using European Quality of Life Five Dimension Five Level Scale Questionnaire | Up to 2 years
  Will assess the impact on quality of life using European Quality of Life Five Dimension Five Level Scale Questionnaire. Will be modeled using mixed effects linear regression. Within-cohort changes will be estimated using linear contrasts of model parameters.

OTHER OUTCOMES:
Scalp thickness | Up to 18 months
  Will assess the IM-SRT on scalp thickness as determined by magnetic resonance imaging evaluations of scalp thickness in the coronal plane before conformal radiation therapy (XRT), at 9 months, and 18 months after XRT in the study group compared to time-matched historical controls of patients. Mixed effects linear regression will be used to jointly model scalp thickness measurements at pre-treatment, 9 months, and 18 months. Potential confounding factors (chemotherapy, smoking history, diabetes) will also be included in the model. The residual variance covariance matrix will be assumed to have a compound-symmetric structure to account for the correlation among repeated measurements. Linear contrasts will be used to compare the change from pre-treatment to 9 months between IM-SRT and conformal therapy patients and to compare the change from pre treatment to 18 months between IM-SRT and conformal therapy patients.

CONTACTS AND LOCATIONS:
Overall Officials: Wenyin Shi, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Niazi M, Russial O, Cappelli L, Miller R, Chen Y, Vakhnenko Y, Liu H, Shi W. Efficacy of scalp-sparing volumetric-modulated arc therapy approach in reducing scalp radiation dose for patients with glioblastoma: a cross-sectional study. Chin Clin Oncol. 2023 Aug;12(4):36. doi: 10.21037/cco-23-15. PMID 37699601
- See also: Sidney Kimmel Cancer Center — https://www.jeffersonhealth.org/clinical-specialties/cancer
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/